CLINICAL TRIAL: NCT04857177
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group, Phase III Clinical Trial To Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of CKD-701 and Lucentis® in Patients With Neovascular(Wet) Age Related Macular Degeneration
Brief Title: A Study To Evaluate CKD-701 and Lucentis® in Patients With Neovascular(Wet) Age Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 177AMD17019
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Neovascular(Wet) Age Related Macular Degeneration
Keywords: Neovascular(wet) Age related Macular Degeneration; CKD-701
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-701 (Experimental): Drug: CKD-701 (proposed ranibizumab biosimilar)
  Interventions: Drug: CKD-701
- Lucentis® (Active Comparator): Drug: Lucentis® (ranibizumab)
  Interventions: Drug: Lucentis®

INTERVENTIONS:
Drug: CKD-701 — CKD-701 (proposed ranibizumab biosimilar) 0.5mg via intravitreal injection every one month during the loading phase, and intervals of one month based on criteria during the PRN phase.
  Arms: CKD-701
Drug: Lucentis® — Lucentis® (ranibizumab) 0.5mg via intravitreal injection every one month during the loading phase, and intervals of one month based on criteria during the PRN phase.
  Arms: Lucentis®

SUMMARY:
This is a multicenter, randomized, double-blind, active-controlled, parallel group, Phase III Clinical Trial To Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of CKD-701 and Lucentis® in Patients with Neovascular(wet) Age related Macular Degeneration

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either CKD-701 or Lucentis®. Investigational Products (IP) (CKD-701 or Lucentis®) will be administered once a month during the loading phase(the first three months), and for the next nine months(PRN phase), administion will be determined based on the PRN administration criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years
2. Presence in the study eye of active subfoveal CNV lesion due to AMD
3. The total lesion size ≤ 12 DA in the study eye
4. The presence of CNV foci of more than 50% of the total lesion area in the study eye
5. The best-corrected visual acuity within a range from 78 to 34 letters (20/32~20/200) measured using the ETDRS chart in the study eye
6. Written informed consent

Exclusion Criteria:

1. Any previous anti-vascular endothelial growth factor(anti-VEGF) treatment to treat neovascular AMD
2. Presence of eye-related inflammation or infection, such as Infectious ophthalmitis, corneal inflammation, conjunctivitis (including scleromalacia), endocular inflammation
3. Any history or clinical basis of disease affecting the retina except age-related macular degeneration(AMD), such as diabetic retinopathy, diabetic macular edema
4. Presence of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, angioid streaks retinopathy or pathologic myopia
5. Patients with macular abnormalities other than age-related macular degeneration (AMD)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a decrease in the best-corrected visual acuity (BCVA) score of 15 or fewer letters at 3 months versus baseline. | Baseline to 3 months

SECONDARY OUTCOMES:
Mean change in the best-corrected visual acuity (BCVA) score from baseline to 3 months, 6 months and 12 months | Baseline, 3 months, 6 months, 12 months
The proportion of patients with a decrease in the best-corrected visual acuity (BCVA) score of 15 or fewer letters at 6 months, 12 months versus baseline | Baseline, 6 months, 12 months
The proportion of patients with an increase in the best-corrected visual acuity (BCVA) score of 15 or more letters at 3 months, 6 months, 12months versus baseline | Baseline, 3 months, 6 months, 12 months
Change in the Central Retinal Thickness(CRT) at 1 months, 3 months, 6 months, 12months versus baseline | Baseline, 1 months, 3 months, 6 months, 12 months
The proportion of patients with the absence of intraretinal fluid and subretinal fluid at 3 months, 6 months, 12months versus baseline | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Gon Yu, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No